CLINICAL TRIAL: NCT04391075
Title: Analgesia in the Second Stage of Labour - With Special Focus on Pudendal Block
Brief Title: Analgesia in the Second Stage of Labour
Acronym: ASL
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Åsa Waldum, Midwife/PhD student, Oslo University Hospital
Other Study IDs: 2016/18884
Record Dates: First submitted 2020-05-12; First posted 2020-05-18 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Childbirth Experience; Urinary Retention; Satisfaction, Personal; Pain, Obstetric
Keywords: Pudendal nerve block; Urine and urination; Anesthetics; Peripheral nervous system agents
MeSH Terms: conditions — Urinary Retention; Personal Satisfaction; Labor Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed: Pudendal nerve block provided
  Interventions: Procedure: Pudendal nerve block
- Not exposed: Pudendal nerve block is NOT provided

INTERVENTIONS:
Procedure: Pudendal nerve block — Pudendal nerve block provided during last fase of delivery
  Groups: Exposed

SUMMARY:
This study investigates efficacy, safety and childbirth experience in women receiving pudendal block during the final stage of delivery. It is an observational study and half of included primarous women recieve a pudendal block.

DETAILED DESCRIPTION:
Pudendal block is used when there is a need to alleviate pain in the final stage of labour:

* From fully dilated cervix to delivery of the child.
* Associated with pain as the foetus rotates and descends through the pelvis.
* End of second stage: the perineum dilates as the child is being born.

Pudendal block is provided by inserting a needle close to the pudendal nerve that runs through the pelvis and innervates the perineal area.Pudendal block is an old and relatively simple method, but not well studied. The main aim is to study pudendal nerve block as pain relief in final stage of labour for primiparous women delivering vaginally.

The investigators aim to investigate whether possible adverse effects may outweigh the positive analgesic effect in the final stage of labour, or the opposite. The ASL (Analgesia in the Second stage of Labour) study may fill knowledge gaps and add important knowledge regarding pain relief during the final stage of childbirth.

ELIGIBILITY:
Inclusion Criteria:

* Norwegian-speaking/reading
* Primiparity
* Single pregnancy
* Vaginal birth
* Cephalic presentation
* ≥37+0
* Age ≥18 years

Exclusion Criteria:

* Transferre from midwifery-led birth unit
* Allergy to local anaesthesia
* Not valid data on pudendal block

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants is selected from 2 delivery units at Oslo Univeristy Hospital (OUH) in Oslo, Norway. OUH is a third referral hospital, the largest Obstetrics Dept. in Norway, and accounting for 1/6 of all deliveries in Norway (9600 deliveries/year).
Sampling Method: Probability Sample
Enrollment: 1007 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Childbirth experience | Responds to questionnaire 4-12 weeks after delivery.
  Childbirth experience questionnaire (CEQ), total score on a scale from 1.0 to 4.0. Higher score means better experience.
Urinary retention | 3 hours
  Urinary retention after delivery defined as inability to void and need for catheterization within 3 hours.

SECONDARY OUTCOMES:
Pain, obstetric | Responds to questionnaire 4-12 weeks after delivery.
  Measured by Visual Analog Scale (VAS). Scale from 0 to 100, higher scpre means more pain.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Flem Jacobsen, PhD, Principal Investigator — Univeristy of Oslo

IPD SHARING:
Plan to Share IPD: Yes
Anonymous individual participant data for the primary outcome measures will be made available on request, when the study is finished. Access to data will be restricted due to sensitive nature of the data, but will be shared if asked for within the anonymous data restriction imposed by the patient consent and ethical body approval.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available on request within 1 year after study completion.
Access Criteria: Data access will be considered on specific request. Requestors wil be required to sign a Data Access Agreement.